CLINICAL TRIAL: NCT06329466
Title: The Effect of Emotional Freedom Technique (EFT) on Pain Intensity and Menstruation Symptoms in High School Students With Primary Dysmenorea: A Single Blind Randomized Control Study
Brief Title: The Effect of Emotional Freedom Technique (EFT) on Pain Intensity and Menstruation Symptoms
Acronym: EFT
Status: Active, not recruiting | Type: Observational
Sponsor: Gulay Coskun (Other)
Collaborators: Mersin University (Other)
Responsible Party: Sponsor-Investigator, Gulay Coskun, MersinU, Mersin University
Organization: Mersin University (Other)
Other Study IDs: 0000-0002-4205-669X
Record Dates: First submitted 2023-06-11; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Dysmenorrhea Primary
Keywords: Dysmenorrhea Primary; Emotional Freedom Techniques (EFT)
MeSH Terms: interventions — Methods; Population Groups

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Observation: Before starting the application to the adolescents in the study (EFT) group, researcher G.C. Fast and easy application steps will be explained with the demonstration method, supported by visual presentations.
  Care will be taken to provide a suitable, clean and airy environment in which the participants will feel comfortable. EFT training and applications will be held during the lunch break so that students do not experience problems such as being late for class or absenteeism. It will be taught in groups of 10-11 people in order to be sure that each participant has learned and to easily confirm the accuracy of the application. Researcher G.C. The participants will be asked to do it to themselves at the same time while they are doing it on themselves to teach the hitting points and application principles.
  Interventions: Other: intervention (EFT) group
- Control: Students in the control group will not receive any intervention during the EFT application. Participants in the control group will have the MAÖKF and MSQ filled before the first session, at the end of the third cycle and at the end of the fourth cycle without the application. In order to eliminate ethical problems that may occur in the control group, EFT application will be taught to the participants in this group after the data collection process of the research is completed.
  Interventions: Other: intervention (EFT) group

INTERVENTIONS:
Other: intervention (EFT) group — It is the group to which EFT is applied.

SUMMARY:
The most important indicator of the fertility period, which has an important place in a woman's life, is the menstrual cycle, which begins with menarche and continues until menopause. In this natural process that takes place every month physiologically, some women experience significant pain [1]. This condition, defined as dysmenorrhea (painful menstruation), is classified in two ways as primary dysmenorrhea (PD) and secondary dysmenorrhea (SD) [2,3]. PD is the most common women's health problem, especially in adolescents and young adults (10-20 years of age) [1,5].

When studies on the incidence and severity of primary dysmenorrhea are examined, the incidence of PD is seen at rates ranging from 40-90% [5-8].

The main goal of the treatment approach to PD, which negatively affects women's quality of life in many ways, is to relieve the woman by reducing the pain. Emotional Freedom Technique (EFT) is one of the non-pharmacological and integrated treatment methods for women with primary dysmenorrhea. This practice, which is also referred to as EFT stroke/touch in most sources, is based on expressing the problem by touching the energy meridian points of the body, as in acupuncture and acupressure.

Considering the results of the studies, it can be said that EFT is effective in the management of pain and the negative effects caused by the restrictions in the life of the person (social and daily living activities, etc.) [27-30]. Thanks to EFT, it is thought that women will contribute to the reduction of the fear and anxiety of experiencing pain just before menstruation and the anxiety that their life will be limited due to this.

Studies investigating the effect of EFT on pain have reported that it is effective in coping with pain [33-35]. However, no randomized controlled study was found in the literature search for the application of EFT in high school students with dysmenorrhea. For this reason, it is thought that if EFT is applied in this age period with a high incidence of dysmenorrhea, important findings can be achieved in terms of parameters such as pain intensity and menstrual symptoms, and it will contribute to the literature by shedding light on similar studies. [36]. Therefore, in this study, it was aimed to determine the effect of the emotional freedom technique applied to high school students with primary dysmenorrhea on pain severity and menstruation symptoms.

DETAILED DESCRIPTION:
Between 26 December 2022 and 26 June 2023, data will be collected from 48 female students who meet the inclusion and exclusion criteria. 9th, 10th and 11th grade female students in the randomized controlled experimental study, whose menstrual pain severity was less than 4, menstrual symptom score was 60 and above, who met all the other inclusion criteria of the study and who declared that they were willing to participate in the study. planned with. Permission approval will also be obtained from the parents of the students who volunteer. Whether or not female students experience primary dysmenorrhea in the study will be determined by the questions in the Determination of Conformity to the Criteria Form (Annex-1), which is the first part of the data collection form.

Purpose and Type of Research The study was planned as a prospective, single-blind randomized controlled experimental study to determine the effect of emotional freedom technique (EFT) on pain level and menstrual symptoms in high school students with primary dysmenorrhea. This randomized controlled trial will be reported according to CONSORT guidelines and registered on ClinicalTrials.gov [37].

The universe of the research; The population of the research will be female students between the ages of 14-17 at secondary schools in Ankara between 26 December 2022 and 25 June 2023.

The sample of the research; The sample of the study will consist of 48 female students aged 14-17 in a secondary school in Ankara between 26 December 2022 and 26 May 2023.

In order to determine the high school where the research will be conducted, public high schools located in the central districts of Ankara will be listed. A high school will be determined by simple random sampling method. The number of female students between the ages of 14-17 studying at the determined high school will be determined by the Stratified Sampling Method according to the class [38].

Location and Features of the Research The research is planned to be carried out in a high school providing secondary education in Ankara. After obtaining the approval of the ethics committee, a list of public high schools located in nine central districts of Ankara Provincial Directorate of National Education (Altındağ, Çankaya, Etimesgut, Gölbaşı, Keçiören, Mamak, Pursaklar, Sincan and Yenimahalle) will be created and a high school will be determined by simple random sampling method. . It is planned to hold an information meeting in the conference hall of the high school to be determined.

Students will be taught the EFT application in the meeting room or empty classroom within the high school. In the first, second and third cycles, students will be able to do their applications at school (lunch break/after school) or at home, by determining the days and hours suitable for them under the control of the researcher.

Identification of Participants In order to determine the participants in the research, an information meeting about the research will be held in the conference hall of the school for female students between the ages of 14-17 who are studying at high school. At the end of the meeting, a list of students who volunteered to participate in the research will be made. These students will be given informed voluntary consent forms for both themselves and their legal representatives to sign. The next day, the signed documents will be taken by going to the school. A Compliance Determination Form will then be applied to identify students who experience primary dysmenorrhea, in other words, pain during menstrual periods. Accordingly, students with a menstrual pain severity of at least 4 according to the Visual Pain Scale, a score of 60 or higher on the Menstruation Symptom Scale, and meeting other selection criteria will be selected for inclusion in the study.

Randomization 48 students from the 9th, 10th and 11th grades of the high school will be included in the study. First of all, the number of students entering each stratum will be determined according to the stratified random sampling method. Then, in the assignment process of the students to be taken from these classes to the experimental and control groups, block randomization will be applied in order to eliminate the selection bias and to keep the number of individuals between the groups in balance.

blinding In the research, EFT will not be blinded as it will be done face to face by the researcher. However, the participants will practice and be blinded without knowing whether they are in the study group or the control group. Thus, the research will be carried out as a single-blind randomized controlled trial. When the research is completed, the data of the study (EFT) and control groups (coded as A or B) will be transferred to the computer environment by an independent researcher, and the data will be analyzed by a statistician and the findings will be reported.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 14-17,
* Willing to participate in the research,
* Open to communication,
* Having opportunities (computer, internet, etc.) to attend trainings online,
* Having a regular menstrual period (occurring at intervals of 21-35 days and lasting 3-8 days),
* Menstrual pain severity is at least 4 according to the Visual Pain Scale,
* A score of 60 or more on the Menstruation Symptom Scale,
* Applying to the obstetrician due to menstrual pain and determined not to have a pathology causing secondary dysmenorrhea,
* Not using hormonal contraception,
* Does not have a systemic and chronic disease,
* EFT will block/limit the application no physical/mental health problems,
* No psychiatric problems
* Female students with primary dysmenorrhea studying in the 9th, 10th and 11th grades.

Exclusion Criteria:

* under 14 years old and over 17 years old,
* Those who do not agree to participate in the research,
* Unable to communicate
* Do not have opportunities (computer, internet, etc.) to attend trainings online,
* Not having a regular menstrual period,
* Menstrual pain severity is less than 4 according to the Visual Pain Scale,
* A score of 59 or less on the Menstruation Symptom Scale,
* Applying to the obstetrician due to menstrual pain and determined to have a pathology causing secondary dysmenorrhea,
* Using hormonal contraception,
* Having a systemic and chronic disease,
* EFT will block/limit the application have physical/mental health problems,
* Having a psychiatric problem,
* 12th grade female students without primary dysmenorrhea.

Ages: 14 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — The female just have dysmenhorea
Study Population: The High School Female students with primary dysmenorrhea
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2022-01-28 (Actual); Primary Completion 2024-06-25 (Estimated); Study Completion 2024-07-25 (Estimated)

PRIMARY OUTCOMES:
Mcgill Pain Scale | Before the study (Pre-test) 2. End of the application (week 12) 3. Post-test (at the end of the 16. week).
  Mcgill Pain Scale Short Form (MAS-SF) The Mcgill Pain Scale Short Form was developed by Ronald Melzack in 1987 to determine the nature, effect, and overall pain intensity of pain [41].
  In the first part of the Mcgill Pain Scale Short Form, there are 15 word groups describing the sensory/perceptual pain dimension (first 11 words) and emotional/emotional pain dimension (last four words).
  In the second part of the scale, the severity of the pain at that moment is determined from the patient by using the VAS.
  In the third part of the scale, a six-point Likert type scale is used to determine the general pain intensity. Scale; It consists of expressive values ranging from 0 = no pain, 1 = mild, 2 = bothersome, 3 = distressing, 4 = terrible, 5 = unbearable pain.
Menstruation Symptom Scale | Before the study (Pre-test) 2. End of the application (week 12) 3. Post-test (at the end of the 16. week).
  Menstruation Symptom Scale (MSI) It was developed by Chesney and Tasto in 1975 to assess menstrual pain and symptoms [43]. The scale, which is a five-point Likert type and consists of 24 items, was updated by Negriff et al. in 2009 by re-evaluating its factor structure and usability. The MSÖ score is calculated by taking the total mean score of the items in the scale. An increase in the mean score indicates an increase in the severity of menstrual symptoms. The score obtained from the sub-dimensions in the scale is calculated by taking the total score average of the items in the sub-dimensions. An increase in the mean score for the sub-dimensions indicates an increase in the severity of menstrual symptoms related to that sub-dimension [45].
  The highest value of the scale is 110 (menstrual problems most) and the lowest value is 22 (menstrual problems least).
VAS pain scale | Pre-Study will be applied to determine compliance with the criteria.
  Visual Analogue Scale (VAS)
  Different scales are used in studies to measure the level of pain. In our study, the pain intensity of the participants will be determined by using the Visual Analogue Scale (VAS) in the Determination of Compliance with the Criteria Form. VAS has been developed in order to be able to specify the severity of pain more easily by converting some values that cannot be measured numerically. VAS is a safe, easily applicable measurement tool that has been generally accepted in the world literature for many years. A low score on the VAS indicates low/low pain intensity, and a high score indicates high/severe pain [39,40].
  The highest value of the scale is 10 (most pain) and the lowest value is 0 (no pain).

CONTACTS AND LOCATIONS:
Overall Officials: Duygu Vefikuluçay Yılmaz, Prof, Study Chair — Mersin University Faculty of Nursing; Gülay Coşkun, Principal Investigator — Mersin University Faculty of Nursing
Locations (1):
- Mersin University, Yenişehir, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No